CLINICAL TRIAL: NCT04555421
Title: Using the Lumen Device for Prediabetes Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Metaflow Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0523-20
Record Dates: First submitted 2020-09-16; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: PreDiabetes; Overweight and Obesity
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumen device usage and diet guidelines (Experimental)
  Interventions: Device: Lumen

INTERVENTIONS:
Device: Lumen — Subjects will use the Lumen device and mobile phone application, which will guide their diet, sleep, and routines according to their Lumen measurements. In addition, a Lumen coach will be assigned to the subjects, and they will have a 30 minutes video call with the coach during the familiarization stage, in order to acquaint them with Lumen and explain them about the application and the nutritional guidance.

SUMMARY:
To examine the effect of using Lumen on metabolic parameters and anthropometric variables. This will be done from baseline to the end of a 12 weeks intervention in adults with prediabetes..

DETAILED DESCRIPTION:
A single arm intervention evaluation for 12 weeks (pre-post analysis) was designed for the study. After initial screening of the subjects, they will be familiarized with Lumen and will learn on how to take a measure. After 2 days of using Lumen device at home for acquaintance and calibration, subjects will arrive to the clinic and several baseline measurements will be taken, including blood samples and anthropometric variables. Then, subjects will use Lumen at home and will take a Lumen measurement each day for a period of 12 weeks. Subjects will take a Lumen measurement each morning at fasted state and will get a nutritional plan according to their result. In addition, subjects will be guided to log in the last time they consumed a meal (how long they fasted for), the duration of their sleep, and if they managed to follow the previous day recommendations. Moreover, the Lumen application will encourage the subjects to take more measurement throughout the day, in particular in response to food intake as well as before and after workouts. Lumen coach will remotely support the subjects via Lumen's mobile phone application and will provide clarifications and guidelines if needed based on the Lumen metric. Finally, subjects will return to the clinic for their final assessment which would include taking blood samples and anthropometric variables again.

The study will include 40 subjects the most with a minimal target of 30 subjects. The number of subjects was determined based on power analysis made according to a study evaluating HbA1c levels in prediabetic subjects who received low-carb diet for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

BMI ≥ 27 to ≤ 40 HbA1c ≥ 5.7% to ≤6.4% Fasting glucose ≥ 100 mg/dl to ≤ 125 mg/dl Not treated with diabetes-related medications

Exclusion Criteria:

Medications:

1. Insulin and medications for glycemic control
2. Antipsychotics
3. Diuretics
4. Anti-retrovirals
5. Corticosteroids
6. Oncologic treatment
7. Thyroid hormones (if endocrinological control is good, can be included).

Conditions:

1. Previous diagnosis of diabetes
2. G6PD deficiency
3. Renal disease
4. Hepatic disease
5. Pregnancy
6. Hematological (anemia)
7. Suffered heart attack, stroke, or transient ischemic attack in the past 6 months
8. Uncontrolled hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure > 105 mm Hg)
9. Treatment of cancer (excluding surgery alone) within the past 2 years (excluding skin cancer)
10. Reported chest pain, shortness of breath with minimal activity or at rest, or unexplained dizziness or fainting with physical activity
11. Chronic lung disease (chronic obstructive pulmonary disease or asthma requiring oxygen therapy)

Personal requirements:

1. Inability to read and understand English
2. Inability to use a smartphone
3. Any issues arise with using the Lumen device and application
4. Aerobic exercise > 3 times per week
5. Active participation in diet counseling or active weight loss (> 3 kg in the past one month)
6. Change of diet or physical activity in the last 3 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Weight change | from baseline to 12 weeks
  % weight change
Fat percentage | from baseline to 12 weeks
  % change in fat percentage

SECONDARY OUTCOMES:
Blood tests changes - glycemic control | from baseline to 12 weeks
  HbA1C (%)
Blood tests changes- lipid panel change | from baseline to 12 weeks
  Triglycerides, HDL and LDL cholesterol, total cholesterol) - change in mg/dl
Blood tests changes - glycemic control | from baseline to 12 weeks
  Fasting glucose (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Endocrinology, Metabolism and Hypertension, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No